CLINICAL TRIAL: NCT07253285
Title: Efficacy, Safety and Pharmacokinetics of Cagrilintide s.c. 2.4 mg as Monotherapy and in Combination With Semaglutide s.c. 2.4 mg (CagriSema) Once Weekly for Weight Management in Chidren and Adolescents With Overweight or Obesity
Brief Title: A Research Study on How Well Cagrilintide and CagriSema Work in Children and Adolescents With Excess Body Weight
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4968; U1111-1299-4751 (Other: World Health Organization (WHO)); 2023-509176-42 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures. The main phase of the study is double blinded and followed by an open label extension phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CagriSema (Experimental): Participants will receive once weekly subcutaneous (s.c.) dose of CagriSema (cagrilintide and semaglutide) in a dose escalation regimen in the main phase for up to 16 weeks and maintained for 52 weeks and further continue to receive the same dose or maximum tolerated dose (MTD) in the open-label extension phase for up to 156 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide; Drug: Placebo cagrilintide; Drug: Placebo semaglutide
- Semaglutide (Experimental): Participants will receive once weekly s.c. dose of semaglutide in a dose escalation regimen in the main phase for up to 16 weeks and maintained for 52 weeks.
  Interventions: Drug: Semaglutide; Drug: Placebo semaglutide
- Cagrilintide (Experimental): Participants will receive once weekly s.c. dose of cagrilintide in a dose escalation regimen in the main phase for up to 16 weeks and maintained for 52 weeks, further continue to receive the same dose as the dose escalation regimen or MTD in the open-label extension phase for up to 156 weeks.
  Interventions: Drug: Cagrilintide; Drug: Placebo cagrilintide
- Placebo (Placebo Comparator): Participants will receive once weekly s.c. dose of placebo matched to cagrilintide/semaglutide in a dose escalation regimen in the main phase for up to 16 weeks and maintained for 52 weeks. Participants will further continue to receive the same dose escalation regimen as CagriSema for 16 weeks, later continue to receive the same dose or MTD in the open-label extension phase for up to 140 weeks.
  Interventions: Drug: Placebo cagrilintide; Drug: Placebo semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive cagrilintide subcutaneously.
  Arms: CagriSema; Cagrilintide
Drug: Semaglutide — Participants will receive semaglutide subcutaneously.
  Arms: CagriSema; Semaglutide
Drug: Placebo cagrilintide — Participants will receive placebo matched to cagrilintide subcutaneously.
  Arms: CagriSema; Cagrilintide; Placebo
Drug: Placebo semaglutide — Participants will receive placebo matched to semaglutide subcutaneously.
  Arms: CagriSema; Placebo; Semaglutide

SUMMARY:
This study will look at how well CagriSema and cagrilintide help children and adolescents with excess body weight lose weight. The study has 2 parts: main and extension study. In the main study, participants will either get CagriSema (a new study drug), cagrilintide (a new study drug), semaglutide (a drug that doctors can already prescribe to adolescents and adults) or placebo (a placebo looks like the treatment being tested, but doesn't have any active ingredients in it). Which treatment participants will get is decided by chance. Participants who get semaglutide in the main study will not take part in the extension study. If participants take part in the extension study, they will get either CagriSema or cagrilintide in this part of the study. Like all drugs, the study drugs may have side effects. The total time participants will be in the main study is about 1 year and 6 months. If participants take part in the extension study, the total time is about 4 years and 10 months.

ELIGIBILITY:
Inclusion criteria:

* Informed consent of parent(s) or legally acceptable representative (LAR) of participant and child assent, as age-appropriate, obtained before any study related activities. Study related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* The parent(s) or LAR of the child must sign and date the Informed Consent Form (according to local requirements)
* The child must sign and date the Child Assent Form or provide oral assent (according to local requirements).
* Male or female.
* Aged 8 to less than (<) 18 years at the time of signing the informed consent.
* Body mass index (BMI), at screening, corresponding to:
* Greater than or equal to (>=) 95th percentile for children aged 8 to < 12 years (Tanner stage 1-5)
* >= 95th percentile or >= 85th percentile with the presence of at least one obesity-related complication including, but not limited to, type 2 diabetes (T2D), hypertension, dyslipidaemia or obstructive sleep apnoea for adolescents aged 12 to < 18 years (Tanner stage 2-5).
* Laboratory parameters, as measured by the central lab at screening, within normal sex- and age-specific ranges of total calcium, phosphate, alkaline phosphatase, parathyroid hormone.
* History of at least one unsuccessful effort to lose sufficient body weight after participation in a structured lifestyle modification programme (diet and exercise counselling) for at least 3 months.
* Body weight greater than (>) 45 kilograms (kg) at screening.

For participants with T2D at screening the following inclusion criteria also apply

* Glycated haemoglobin (HbA1c) less than or equal to (<=)10.0 percent (%) (86 millimoles per mole [mmol/mol]) as measured by central laboratory at screening.
* Treatment with lifestyle intervention or treatment with metformin according to local label.
* Treatment with metformin should be stable (same dose and dosing frequency) for at least 56 days before screening.

Key exclusion criteria:

* Treatment with any medication prescribed for obesity or weight management within 90 days before screening.
* Previous or planned (during the study period) obesity treatment with surgery or a weight loss device. However, the following are allowed:
* Liposuction and/or abdominoplasty, if performed > 1 year before screening.
* Adjustable gastric banding, if the band has been removed > 1 year before screening.
* Intragastric balloon, if the balloon has been removed > 1 year before screening.
* Duodenal-jejunal bypass liner (e.g., Endobarrier), if the sleeve has been removed >1 year before screening.
* Uncontrolled thyroid disease.
* Endocrine, hypothalamic, or syndromic obesity.
* A self-reported (or by parent(s)/LAR, where applicable) change in body weight > 5 % within 90 days before screening irrespective of medical records.
* Type 1 diabetes or monogenic diabetes. For participants without T2D at screening the following exclusion criteria also apply
* HbA1c greater than or equal to 6.5% (48 mmol/mol) as measured by the central laboratory at screening.
* Treatment with glucose-lowering agent(s) prescribed for the indication of diabetes or pre-diabetes within 90 days before screening.

For participants with T2D at screening the following exclusion criteria also apply

* Known hypoglycaemic unawareness as indicated by the investigator according to Clarke's questionnaire.
* Recurrent severe hypoglycaemic episodes within 1 year before screening, as judged by the investigator.
* Positive insulinoma associated protein-2 (IA-2) antibodies or anti-glutamic acid decarboxylase (anti-GAD) antibodies.
* Treatment with any medication for the indication of diabetes other than those stated in the inclusion criteria within 90 days before screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 460 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2030-03-20 (Estimated); Study Completion 2033-09-20 (Estimated)

PRIMARY OUTCOMES:
Relative change in body mass index (BMI) | Baseline (week 0), week 68
  Measured in percentage (%).

SECONDARY OUTCOMES:
Relative change in body weight | Baseline (week 0), week 68
  Measured in %.
Change in BMI Standard Deviation Score (SDS) | Baseline (week 0), week 68
  Measured as SDS score.
Relative change in BMI | Baseline (week 0), week 68 and week 224
  Measured in %.
Number of participants in weight category reduction | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved greater than or equal to (>=) 5 percent (%) reduction of body weight (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=10% reduction of body weight (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=15% reduction of body weight (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=20% reduction of body weight (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=25% reduction of body weight (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=5% reduction of BMI (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=10% reduction of BMI (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=15% reduction of BMI (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=20% reduction of BMI (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved >=25% reduction of BMI (yes/no) | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who achieved normal BMI | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants who shifted from obese to non-obese BMI class | Baseline (week 0), week 68
  Measured as count of participants.
Change in waist circumference | Baseline (week 0), week 68 and week 224
  Measured in centimeter (cm).
Change in waist-to-height ratio | Baseline (week 0), week 68
  Measured as ratio.
Absolute change in total fat mass by dual energy X-ray absorption (DXA) | Baseline (week 0), week 68
  Measured in kilograms (kg).
Relative to baseline change in total fat mass by DXA | Baseline (week 0), week 68
  Measured in %.
Relative to total body mass change in total fat mass by DXA | Baseline (week 0), week 68
  Measured in % points.
Absolute change in visceral fat mass by DXA | Baseline (week 0), week 68
  Measured in kg.
Relative to baseline change in visceral fat mass by DXA | Baseline (week 0), week 68
  Measured in %.
Relative to total body mass change in visceral fat mass by DXA | Baseline (week 0), week 68
  Measured in % points.
Absolute change in lean body mass by DXA | Baseline (week 0), week 68
  Measured in kg.
Relative to total body mass change in lean body mass by DXA | Baseline (week 0), week 68
  Measured in % points.
Absolute change in total (neck-to-knee) muscle and fat volumes by Magnetic Resonance Imaging (MRI) - total muscle and total fat | Baseline (week 0), week 68 and week 224
  Measured in liters (L).
Relative to baseline change in total (neck-to-knee) muscle and fat volumes by MRI - total muscle and total fat | Baseline (week 0), week 68 and week 224
  Measured in %.
Change in ectopic fat content by MRI - liver fat MRI-Proton Density Fat Fraction (MRI-PDFF), pancreatic fat, kidney fat and thigh muscle fat infiltration | Baseline (week 0), week 68 and week 224
  Measured in % points.
Absolute change in abdominal fat volumes by MRI - subcutaneous fat and visceral fat | Baseline (week 0), week 68 and week 224
  Measured in liters.
Relative to baseline change in abdominal fat volumes by MRI - subcutaneous fat and visceral fat | Baseline (week 0), week 68 and week 224
  Measured in %.
Absolute change in thigh muscle and fat volumes by MRI - thigh fat free muscle and thigh subcutaneous fat | Baseline (week 0), week 68 and week 224
  Measured in liters.
Relative to baseline change in thigh muscle and fat volumes by MRI - thigh fat free muscle and thigh subcutaneous fat | Baseline (week 0), week 68 and week 224
  Measured in %.
Ratio to baseline in liver stiffness measured by Magnetic Resonance Elastography (MRE) | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Change in BMI percentage of the 95th percentile | Baseline (week 0), week 68
  Measured in % points.
Ratio to baseline highly sensitive C-reactive protein (hs-CRP) | Baseline (week 0), week 68
  Measured as ratio.
Ratio to baseline in lipids: Total cholesterol | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Ratio to baseline in lipids: High Density Lipoprotein (HDL) cholesterol | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Ratio to baseline in lipids: Low Density Lipoprotein (LDL) cholesterol | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Ratio to baseline in lipids: Very Low Density Lipoprotein (VLDL) cholesterol | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Ratio to baseline in lipids: Triglycerides | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Ratio to baseline in lipids: Non-HDL cholesterol | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Change in Alanine Transaminase (ALT) | Baseline (week 0), week 68 and week 224
  Measured in Units per Liter (U/L).
Change in systolic blood pressure | Baseline (week 0), week 68 and week 224
  Measured in millimeters of mercury (mmHg).
Change in diastolic blood pressure | Baseline (week 0), week 68 and week 224
  Measured in mmHg.
Ratio to baseline in liver stiffness measured by ultrasonographic methods | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Change in glycated haemoglobin (HbA1c) (% points) | Baseline (week 0), week 68 and week 224
  Measured in % points.
Change in HbA1c (millimoles per mole [mmol/mol]) | Baseline (week 0), week 68 and week 224
  Measured in mmol/mol.
Change in Fasting Plasma Glucose (FPG) (millimoles per liter [mmol/L]) | Baseline (week 0), week 68
  Measured in mmol/L.
Change in FPG (milligrams per deciliter [mg/dL]) | Baseline (week 0), week 68
  Measured in mg/dL.
Ratio to baseline in fasting serum insulin | Baseline (week 0), week 68 and week 224
  Measured as ratio.
Number of participants with prediabetes who achieved HbA1c less than (<) 5.7% (defined as 5.7 % less than or equal to [<=] HbA1c <6.5 %) at baseline | At week 68
  Measured as count of participants.
Number of participants with normoglycemia (defined as HbA1c < 5.7 %) at baseline, development of HbA1c greater than or equal to (>=) 5.7 % | At week 68
  Measured as count of participants.
Number of participants with prediabetes (5.7 % <= HbA1c < 6.5 %) at baseline, development of HbA1c >= 6.5% | At week 68
  Measured as count of participants.
Number of participants with HbA1c >=6.5% at baseline, achievement of HbA1c <6.5% | At week 68
  Measured as count of participants.
Number of participants taking glucose lowering medication at baseline, stop or decrease | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants taking antihypertensive medication at baseline, stop or decrease | Baseline (week 0), week 68
  Measured as count of participants.
Number of participants taking lipid lowering medication at baseline, stop or decrease | Baseline (week 0), week 68
  Measured as count of participants.
Impact of Weight on Quality of Life-Kids (IWQOL Kids) - Physical comfort domain score | Baseline (week 0), week 68 and week 224
  Measured as score points. IWQOL-Kids measures weight-related quality of life in adolescents (ages 11-19 years) but will be administered to all study participants. The measure consists of 27-items yielding 4 sub-scale scores, and 1 total score. Higher scores indicate better weight-related quality of life. Subscale scores (score range): physical comfort (0-100), body esteem (0-100), social life (0-100), family relations (0-100) and total score (0-100).
IWQOL Kids - Body esteem domain score | Baseline (week 0), week 68 and week 224
  Measured as score points. IWQOL-Kids measures weight-related quality of life in adolescents (ages 11-19 years) but will be administered to all study participants. The measure consists of 27-items yielding 4 sub-scale scores, and 1 total score. Higher scores indicate better weight-related quality of life. Subscale scores (score range): physical comfort (0-100), body esteem (0-100), social life (0-100), family relations (0-100) and total score (0-100).
IWQOL Kids - Social life domain score | Baseline (week 0), week 68 and week 224
  Measured as score points. IWQOL-Kids measures weight-related quality of life in adolescents (ages 11-19 years) but will be administered to all study participants. The measure consists of 27-items yielding 4 sub-scale scores, and 1 total score. Higher scores indicate better weight-related quality of life. Subscale scores (score range): physical comfort (0-100), body esteem (0-100), social life (0-100), family relations (0-100) and total score (0-100).
IWQOL Kids - Family-relations score | Baseline (week 0), week 68 and week 224
  Measured as score points. IWQOL-Kids measures weight-related quality of life in adolescents (ages 11-19 years) but will be administered to all study participants. The measure consists of 27-items yielding 4 sub-scale scores, and 1 total score. Higher scores indicate better weight-related quality of life. Subscale scores (score range): physical comfort (0-100), body esteem (0-100), social life (0-100), family relations (0-100) and total score (0-100).
IWQOL Kids - Total score | Baseline (week 0), week 68 and week 224
  Measured as score points. IWQOL-Kids measures weight-related quality of life in adolescents (ages 11-19 years) but will be administered to all study participants. The measure consists of 27-items yielding 4 sub-scale scores, and 1 total score. Higher scores indicate better weight-related quality of life. Subscale scores (score range): physical comfort (0-100), body esteem (0-100), social life (0-100), family relations (0-100) and total score (0-100).
Control of Eating Questionnaire (COEQ) | Baseline (week 0), week 68 and week 224
  Measured as score points. CoEQ is a 19-item multidimensional patient reported outcome (PRO) that assesses the experience of hunger, satiety, and severity and type of food cravings. CoEQ consists of 4 subscales that measure craving control (5 items), positive mood (4 items), craving for sweet (4 items), craving for savoury food (4 items), and 2 single items that address hunger and satiety. Each item is evaluated on a 0-10 (i.e., 11-point) numeric rating scale. The total score for each subscale is calculated as the sum of the item scores divided by the number of items in the subscale. Scores ranges are thus: Craving Control 0-50/5 = 0-10); Positive Mood (0-40/4 = 0-10); Craving Sweet (0-40/4 = 0-10); Craving Savoury food (0-40/4 = 0-10); single items that address hunger and satiety (0-10). For the craving control subscale, the subscale score is reversed so that a higher score represents a greater level of craving control.
Change in proteomics-based serum biomarkers including biomarkers for metabolic dysfunction-associated steatohepatitis (MASH) | Baseline (week 0), week 68 and week 224
  Measured as counts.
Number of treatment-emergent adverse events (TEAEs) | Baseline (week 0), week 68 and week 224
  Measured as count of events.
Number of treatment-emergent serious adverse events (TESAEs) | Baseline (week 0), week 68 and week 224
  Measured as count of events.
Number of treatment-emergent hypoglycaemic episodes | Baseline (week 0), week 68 and week 224
  Measured as count of events.
Change in pulse rate | Baseline (week 0), week 68
  Measured in beats per minute (beats/min).
Change in calcitonin | Baseline (week 0), week 68
  Measured in nanograms per liter (ng/L).
Apparent clearance (CL/F) of semaglutide and cagrilintide at steady state | Baseline (week 0), week 68
  Measured in liters per hour (L/h).
Average concentration (Cavg) of semaglutide and cagrilintide at steady state | Baseline (week 0), week 68
  Measured in nanomoles per liter (nmol/L).
Area under the steady-state concentration-time curves (AUCt) in the dosing interval of semaglutide and cagrilintide | Baseline (week 0), week 68
  Measured in hours nanomoles per liter (h·nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (116):
- United States (33):
  - Neighborhood Healthcare, Escondido, California
  - Encore Medical Research LLC, Hollywood, Florida
  - Jacksonville Ctr for Clin Res, Jacksonville, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Columbus Research Foundation, Columbus, Georgia
  - Accel Research Sites-NeuroStudies, Decatur, Georgia
  - Eastside Bariatric and Gen Surg, Snellville, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - IU Health - Riley Physicians Endo-Diab, Indianapolis, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Pennington Biomed Res Ctr, Baton Rouge, Louisiana
  - Barry J. Reiner, MD LLC, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - AES Minneapolis DRS, Richfield, Minnesota
  - UBMD Physicians Group - Pediatrics - Conventus, Buffalo, New York
  - SUNY Upstate Medical Univ - Syracuse, Syracuse, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - Centricity Research - Ohio, Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Children's Physicians OU, Oklahoma City, Oklahoma
  - UPMC Child Hosp-Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health-Ped Endo, Greenville, South Carolina
  - Coastal Carolina Research Ctr, North Charleston, South Carolina
  - Monument Health Clinical Rsrch, Rapid City, South Dakota
  - LifeDoc Health, Memphis, Tennessee
  - DM Clinical, Houston, Texas
  - DM Clinical, San Antonio, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Consano Clin Res-Shavano Park, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Wee Care Pediatrics, Syracuse, Utah
- Australia (3):
  - Westmead Children's Hospital- The Clinical Research Centre, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's' Hospital, Nedlands, Western Australia
- Austria (2):
  - Universitätsklinik Kinder-Jugendheilkunde Innsbruck, Innsbruck
  - Universitätsklinik für Kinder und Jugendheilkunde Haus E, Salzburg
- Belgium (2):
  - UZ Brussel - Universitair Ziekenhuis Brussel, Brussels
  - UZA - UZ Antwerpen - Kinderziekenhuis, Edegem
- Bulgaria (4):
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Pediatrics, Plovdiv
  - SHATPD - Prof. Ivan Mitev EAD, Sofia
  - Medical center Children's Health EOOD, Sofia
  - UMHAT Sveta Marina EAD, First Pediatric Clinic, Varna
- China (9):
  - Capital Center for Children's Health, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Wuhan Children Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Bethune Hospital of Jilin University-Pediatric, Changchun, Jilin
  - Shandong Provincial Hospital-Pediatric, Jinan, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
- Colombia (2):
  - Servicios de Salud Ips Suramericana S.A.S., Medellín, Antioquia
  - Fundación Santa Fe de Bogotá, Bogotá
- Croatia (3):
  - Clinical Hospital Centre Rijeka_Pediatric, Rijeka
  - KBC "Sestre Milosrdnice", Zagreb
  - Klinika Za Djecje Bolesti Zagreb_Pediatric department, Zagreb
- Denmark (2):
  - Aalborg Universitetshospital - Børne og Ungeafdelingen, Aalborg
  - Holbæk Sygehus - Børne- og Ungeafdelingen, Holbæk
- Hungary (3):
  - Észak-Közép-budai Centrum, Szent János Kórház és Szakrendelő, Budapest
  - Semmelweis Egyetem ÁOK, Budapest
  - Szegedi Tudományegyetem Gyermekgyógyászati Klinika, Szeged
- India (9):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - BAPS Pramukh Swami Hospital, Surat, Gujarat
  - Indira Gandhi Institute of child health, Bangalore, Karnataka
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Maulana Azad Medical College, Delhi, New Delhi
  - Regency Hospital, Kanpur, Uttar Pradesh
  - Institute of Child Health, Kolkata, West Bengal
  - Excel Endocrine Centre, Kolhāpur
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Israel (3):
  - Rambam MC - Department of Pediatrics A, Haifa
  - Schneider MC - Endrocrinology and Diabetes, Petah Tikva
  - Shamir MC - Pediatric and Adolescents Endocrinology unit, Ẕerifin
- Italy (4):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico - UO Endocrinologia, Milan, Lombardy
  - AOU Maggiore della Carità di Novara - Dipartimento Interaziendale Strutturale Materno Infantile - SCDU Pediatria, Novara, Piedmont
  - IRCCS materno infantile Burlo Garofolo - Clinica Pediatrica, Trieste
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Civile Maggiore Borgo Trento, Verona
- Malaysia (3):
  - Hospital Tunku Azizah, Kampung Baru, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Sibu, Sibu, Sarawak
- Mexico (3):
  - CHRISTUS - Latam Hub Excellence and Innovation Center, Monterrey, Nuevo León
  - IECSI Centro de Investigación Clínica, Monterrey, Nuevo León
  - Consultorio de Endocrinología y Pediatría, Puebla City
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Meander Medisch Centrum, Amersfoort
- Poland (4):
  - Samodzielny Zespół Publicznych Zakładów Opieki Zdrowotnej im. Dzieci Warszawy w Dziekanowie Leśnym, Dziekanów Leśny
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Szyszko, Zabrze
- Portugal (3):
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - Hospital CUF Porto S.A., Porto
  - Unidade Local De Saude De Gaia/Espinho E.P.E., Vila Nova de Gaia
- Romania (4):
  - Spitalul Judetean de Urgenta Dr. Constantin Opris Baia Mare, Baia Mare
  - Kilostop Junior SRL, Bucharest
  - Spitalul Clinic de Urgenta pentru Copii "M.S.Curie", Bucharest
  - Spitalul Clinic Judetean De Urgenta Pius Brinzeu Timisoara, Timișoara
- Serbia (3):
  - University Children's Hospital Tirsova, Belgrade
  - Institute for Mother and Child Health Care of Serbia, Belgrade
  - Institute for Health Care of Children and Adolescents, Novi Sad
- Slovakia (3):
  - Narodny Ustav Detskych Chorob, Bratislava
  - Detska Fakultna nemocnica Kosice, Košice
  - Narodny Endokrinologicky a diabetologicky ustav, Ľubochňa
- Spain (3):
  - Hospital Vall d'Hebrón_Endocrinología pediatríca, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitario Virgen del Rocío, Seville
- Sweden (2):
  - Barn och ungdomscentrum Västerbotten, Umeå
  - Uppsala universitetssjukhus, Uppsala
- Taiwan (2):
  - Taipei Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Thailand (2):
  - King Chulalongkorn Memorial Hospital_Ped-Nutrition, Bangkok
  - Thammasat Hospital_CRC, Pathum Thani
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Alder Hey Children's Hospital, Liverpool
  - University College Hospital - Paediatric Services, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on NovoNordisk trials.com.
URL: https://novonordisk-trials.com